CLINICAL TRIAL: NCT00099528
Title: REN-1654 in Post-Herpetic Neuralgia: a Multi-Center, Placebo Controlled, 3-week Dose-Finding Study, With a 3-Week Active-Treatment Extension
Brief Title: Dose-Finding Study of REN-1654 in Patients With Post-Herpetic Neuralgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Renovis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REN-1654-2-02
Record Dates: First submitted 2004-12-15; First posted 2004-12-16 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2005-03

CONDITIONS: Neuralgia; Shingles; Peripheral Nervous System Disease
Keywords: Post-herpetic neuralgia; Shingles; Herpes Zoster; Neuropathic pain; Neuralgia; Anti-TNF agents; Inflammatory cytokines; Hyperalgesia; Allodynia; Irritable nociceptor
MeSH Terms: conditions — Neuralgia; Herpes Zoster; Peripheral Nervous System Diseases; Neuralgia, Postherpetic; Hyperalgesia

INTERVENTIONS:
Drug: REN-1654

SUMMARY:
The purpose of this study is to gain initial safety and efficacy data on the experimental agent REN-1654 in patients with painful post-herpetic neuralgia (PHN).

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized, placebo-controlled, dose-finding study. After screening and baseline clinical assessments, subjects will be randomly assigned to receive 30 or 100 mg REN-1654 by mouth (p.o.), or matching placebo, once daily for 3 weeks. After 3 weeks of treatment, the clinical assessments will be repeated. Subjects who complete the 3 week placebo-controlled segment may enter the 3-week active-treatment extension segment, during which subjects in the REN-1654 30 mg group will remain on that dose, subjects who were given placebo in the previous segment will receive REN-1654 100 mg daily, and subjects who received REN 1654 100 mg in the first 3 week study segment will discontinue dosing. Double-blind conditions will be maintained through the placebo-controlled active treatment period (primary efficacy endpoint) and for those continuing dosing into the 3-week second active treatment period. The clinical assessments will be repeated at the end of 6 weeks, after which all subjects will discontinue treatment and return 2 weeks later for the final clinical assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, aged 55 years or older, able and willing to provide written informed consent to participate in the study.
2. Able to read, understand and follow the study instructions, including completion of pain intensity rating scales.
3. History of herpes zoster cutaneous rash, followed by persistent pain for 2 to 18 months after the onset of the rash until the time of dosing with study medication.
4. A screening Daily Spontaneous Pain Rating (for the prior 24-hour period) of at least 4, using an 11-point categorical pain intensity scale with 0 as "no pain" and 10 as "the worst pain imaginable".
5. A positive (non-zero) Evoked Allodynia score reported at the time of screening using the categorical pain intensity scale in response to at least one of two stimuli: light stroking with a foam brush, or #14 von Frey hair stimulation.
6. Subjects who are compliant in maintaining a Pain Diary between the screening and baseline visits, and who record a Daily Spontaneous Pain Rating score of 4 or greater on at least 3 days during the week prior to the baseline visit.
7. Subjects who at screening are taking analgesics, antidepressants, anticonvulsants, anxiolytics, or muscle relaxants, must have been on each such medication for 4 weeks, and at stable doses for 2 weeks prior to the baseline visit, and must be maintained on the same doses throughout the study.
8. Subjects who at screening are receiving adjunctive analgesic therapy such as acupuncture or biofeedback should either discontinue it or establish a schedule of treatments that will remain consistent for 2 weeks prior to the baseline visit, and throughout the study.
9. Subjects who agree to discontinue topical pain treatments at least 2 weeks before the baseline visit, and agree not to use them during the study.
10. Subjects who agree that they will not receive local, regional or spinal (articular, epidural, or intrathecal) injections of medication for pain treatments within 2 weeks prior to the baseline visit and through the end of the study.
11. If female, must be post-menopausal, surgically sterile, not currently pregnant (verified by a screening pregnancy test) or nursing, and using a reliable contraception method such as intrauterine device (IUD), hormonal birth control pills, or double-barrier method (male condom, female condom or diaphragm with spermicidal jelly).
12. If male, must agree to use double-barrier methods of contraception.

Exclusion Criteria:

1. History of peripheral neuropathy or any chronic pain condition other than PHN.
2. History of hepatic, cardiovascular, renal, gastrointestinal, hematological, neurological, endocrine (including diabetes), metabolic, pulmonary, immunologic (including HIV) or psychiatric disease that in the opinion of the Investigator would pose a significant safety risk for a subject exposed to an investigational compound such as REN-1654, or could significantly diminish the quality of the efficacy data to be collected in the study.
3. History of the following ophthalmic disorders based upon medical review at the screening visit. Subjects will further undergo a screening ophthalmologic assessment. Should any of the following be identified at the screening ophthalmologic examination, the subject will be excluded from the study.

   * Symptomatic cataract, resulting in any visual impairment (if a subject has been diagnosed with cataract to a degree that the cataract interferes with daily living and/or regarding which an ophthalmologist has recommended cataract surgery);
   * Other vision-impairing disorders (if a subject is aware of any eye disorder that has impaired vision, such as age-related macular degeneration, lazy eye (amblyopia), double vision or any optic nerve inflammation); presbyopia and other non-pathological visual acuity deficits are not exclusionary;
   * Herpes zoster ophthalmicus involving the eyeball (if a subject has a history of herpes zoster ophthalmicus causing inflammation of any part of the eye [conjunctiva, cornea, iris, retina, optic nerve]; subjects who only had cutaneous herpes zoster involvement of the eyelid without involvement of the eye may be eligible for the study).
   * Glaucoma or history of ocular hypertension (intraocular pressures greater than 21 mm Hg).
4. Cognitive or psychiatric disorders that may diminish compliance with study procedures, including maintenance of a daily pain diary and accurate dosing of study medication.
5. Screening liver enzyme results greater than the upper limit of the normal range (a value less than one multiple above the upper limit of normal may be acceptable, if approved by the Sponsor before enrollment of the subject).
6. Serum creatinine ≥ 2 mg/dL at screening
7. Use of chemotherapy agents or history of cancer, other than non-metastatic skin cancer that has been completely excised, within five years prior to the screening visit.
8. History of drug or alcohol abuse within one year prior to screening.
9. Use within 2 weeks before start of study investigational compound dosing at baseline and through the end of the study of any investigational compound, any epidural or intrathecal agent, corticosteroid, antiretroviral, etanercept or other anti-TNF-α agent, topical anesthetics, or topical analgesics.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2003-08; Study Completion 2004-12

PRIMARY OUTCOMES:
Change from baseline of the Daily Spontaneous Pain Rating in the most painful area identified at baseline and screening.

SECONDARY OUTCOMES:
(1) Daily Allodynia Rating
(2) Daily Functional Interference Rating for general activity and sleep
(3) Pain Relief Rating (recorded at study visits)
(4) Neuropathic Pain Rating (recorded at study visits)
(5) Evoked Allodynia Rating (recorded at study visits)

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Moreadith, MD, PhD, Study Director — Chief Medical Officer, Renovis, Inc.
Locations (16):
- United States (16):
  - North Alabama Neuroscience Research Associates, Huntsville, Alabama
  - Pivotal Research Centers, Peoria, Arizona
  - HOPE Research Institute, Phoenix, Arizona
  - Advanced Clinical Therapeutics, LLC, Tuscon, Arizona
  - UCSD Center for Pain and Palliative Medicine, La Jolla, California
  - Neurophysiologic Laboratory, Laguna Hills, California
  - Colorado Neurology and Headache Center, Denver, Colorado
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health Center, Dept. Anesthesiology, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - A and A Pain Institute, St Louis, Missouri
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Diagnostic Center of Houston, Houston, Texas
  - University of Wisconsin at Madison, Madison, Wisconsin

REFERENCES:
- See also: Click here for useful information on shingles — http://www.massgeneral.org/conditions/condition.aspx?ID=428&type=conditions